CLINICAL TRIAL: NCT03657862
Title: Comparative Study on the Outcomes of Restoring Untreated and SDF-treated Dentine Caries Lesions in Primary Teeth of Preschool Children
Brief Title: Outcomes of Restoring Untreated and SDF-treated Dentine Caries Lesions in Primary Teeth of Preschool Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW 17-180
Record Dates: First submitted 2018-08-29; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Dental Restoration Failure of Marginal Integrity

STUDY DESIGN:
Intervention Model Description: There are 2 groups of study participants in this study.
  Children with decayed teeth were randomly allocated into either Group 1 (receive topical application of a SDF solution) or Group 2 (placebo) using random numbers, around 10 weeks before receiving dental restoration.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participants (children) did not know their group allocation because a placebo was applied if SDF was not applied.
  The care providers (operator) and the examiners (outcome assessor) were not informed of the children's group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDF treated (Experimental): application of 38% silver diamine fluoride solution
  Interventions: Device: application of 38% silver diamine fluoride solution
- Placebo (Placebo Comparator): application of a placebo (tonic water)
  Interventions: Other: application of a placebo (tonic water)

INTERVENTIONS:
Device: application of 38% silver diamine fluoride solution — SDF solution was painted onto the surface of the carious lesion of the tooth
  Arms: SDF treated
Other: application of a placebo (tonic water) — tonic water was painted onto the surface of the carious lesion of the tooth
  Arms: Placebo

SUMMARY:
The primary objective of this proposed clinical study is to compare the success rates of ART restorations placed in untreated and SDF-treated dentine caries lesions in primary teeth. The secondary objective is to describe the change in parents' satisfaction with the aesthetics of their child's teeth and the change in oral health-related quality of life of preschool children before and after placement of ART restorations.

The study population is preschool children attending kindergartens in different districts in Hong Kong. Children attending grades 1 or 2 in nine kindergartens were invited to receive a free dental examination and had their decayed primary teeth restored, if possible, in the kindergarten by dentists. Parental informed consent was obtained before the dental examination and treatment. Half of the children with decayed primary teeth needing restorations were assigned randomly to receive SDF treatment around 10 weeks before receiving the restoration. The restored teeth were re-examined every 6 months for 24 months to assess the treatment outcome. Parents of the study children were asked to complete a questionnaire at baseline, 6 months and 24 months so as to obtain data on their satisfaction with the aesthetics of their child's teeth and the oral health-related quality of life of the study children.

DETAILED DESCRIPTION:
The study population of this proposed study is Hong Kong preschool children. Children attending grade 1 or 2 in nine selected kindergartens were invited to join this study. An invitation letter with information on the purpose and procedures of the study was sent to the parents of the children through the kindergarten. The parents were asked to give written consent for allowing their child to receive a free oral examination and ART restorations, if indicated for treating the decayed primary teeth in their child's mouth, provided by dentists in the kindergarten. Parental consent were obtained before inclusion of a child in this study.

Cavitated caries lesions in the primary teeth of the study children were restored following the ART procedures (Holmgren et al., 2013). The instruments used were LED illuminated dental mirror, sickle probe, tweezers, hatchet, excavators and flat plastic. The dental restorative material used was a high-strength chemical-cured glass ionomer (Ketac-molar, 3M ESPE, Germany).

At the baseline, all children with parental consent were clinically examined in the kindergarten. Disposable dental mirror attached to a handle with an intra-oral LED light and a ball-ended probe was used. The status of each tooth was recorded. Children who had at least one decayed primary tooth with a cavity into dentine were included into the study. All decayed teeth in the children were restored, except those with inadequate access and those with signs of pulpal pathology. The decayed teeth in half of the children received topical application of a SDF solution (Saforide, Toyo Chemical, Japan), through simple random allocation on a child basis using random numbers, around 10 weeks before receiving the restoration. The time used for placement of each restoration was recorded to the nearest minute.

The children were examined at 6 and will be examined at 12, 18 and 24 months after placement of ART restorations by calibrated examiners who were not involved in the placement of the restorations. The same instruments used in the baseline examination were used in the follow-up examinations. The status of the restorations and restored teeth were assessed and recorded using codes and criteria commonly adopted in previous clinical studies of ART restorations (Lo et al., 2007).

At baseline, information on the children's oral hygiene practice, snacking habit, oral health related quality of life, and parental satisfaction with the appearance of their child's teeth was collected by a self-completed questionnaire. A validated tool for measuring oral health related quality of life of preschool children in Hong Kong, Chinese version of Early Childhood Oral Health Impact Scale (ECOHIS), was used (Lee et al., 2009). The same measurement tool was used at the 6-month and will be used at 24-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy children who had at least one decayed primary tooth with a cavity into dentine

Exclusion Criteria:

* children with serious systemic diseases/conditions or who were uncooperative during treatment
* teeth with signs of pulpal pathology such as having an abscess or discoloured
* caries lesions which did not have adequate access for hand instruments to prepare the cavity for a filling and those that were treated with SDF solution but with most parts still being active

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 195 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
success of the ART restorations | 24 months
  A restoration is classified as success when it is retained on the tooth without major defects or wear and has no associated active caries.

SECONDARY OUTCOMES:
parental satisfaction with aesthetics of their child's teeth as reported in the parent's answer to a question on their satisfaction with the appearance of their child's teeth | 24 months
  parent's answer to a question on their satisfaction with the appearance of their child's teeth. The question is "How satisfied are you with the overall appearance of your child's teeth?" The answer option is a 5-point scale with 5 being very satisfied, 4 being satisfied, 3 being neutral, 2 being dissatisfied, and 1 being very dissatisfied.
oral health related quality of life of the child as assessed by the Early Childhood Oral Health Impact Scale | 24 months
  parents' answers to a series of questions in the Early Childhood Oral Health Impact Scale. This scale contains 13 self-completed questions on various aspects of the impact of child oral health on the daily activities of the child or the family. The answer in each question is on a 5-point scale with 0 being no impact and 4 being great impact. The scale score is the summation of the answer scores to the 13, which can range from 0 to 52. The higher the scale score, the more impacts of oral health on life activities and thus lower quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holmgren CJ, Roux D, Domejean S. Minimal intervention dentistry: part 5. Atraumatic restorative treatment (ART)--a minimum intervention and minimally invasive approach for the management of dental caries. Br Dent J. 2013 Jan;214(1):11-8. doi: 10.1038/sj.bdj.2012.1175. PMID 23306489
- [Background] Lo EC, Holmgren CJ, Hu D, van Palenstein Helderman W. Six-year follow up of atraumatic restorative treatment restorations placed in Chinese school children. Community Dent Oral Epidemiol. 2007 Oct;35(5):387-92. doi: 10.1111/j.1600-0528.2006.00342.x. PMID 17822487
- [Background] Lee GH, McGrath C, Yiu CK, King NM. Translation and validation of a Chinese language version of the Early Childhood Oral Health Impact Scale (ECOHIS). Int J Paediatr Dent. 2009 Nov;19(6):399-405. doi: 10.1111/j.1365-263X.2009.01000.x. PMID 19811551

DOCUMENTS (1):
  • Study Protocol (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT03657862/Prot_000.pdf